CLINICAL TRIAL: NCT06903689
Title: Exploring the Potential Effect of Pentoxifylline in Mitigating Vascular Calcification in Chronic Kidney Disease Patients
Brief Title: Pentoxifylline for Vascular Calcification in Kidney Disease
Acronym: PTX-CALC-CKD
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Dina Massoud Gaber, Resident in Nephrology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS.24.09.2905
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Disease; Vascular Calcification; Kidney Failure, Chronic
Keywords: Kidney Failure, Chronic; Vascular Calcification; Pentoxifylline; CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic; Vascular Calcification; Kidney Failure, Chronic | interventions — Pentoxifylline; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pentoxifylline Arm (Experimental): Participants in this arm will receive Pentoxifylline 400 mg twice daily orally with food, in addition to their conventional medications for chronic kidney disease (CKD). Pentoxifylline treatment will be administered for 6 months, concurrent with the study duration. Conventional medications will continue as prescribed by their treating physician and will be consistent with standard of care for CKD.
  Interventions: Drug: Pentoxifylline 400 MG Oral Tablet
- Conventional Medication Group (Active Comparator): Participants in this arm will receive conventional medications for chronic kidney disease (CKD) only. They will not receive Pentoxifylline. Conventional medications will be administered as prescribed by their treating physician and will be consistent with standard of care for CKD. This arm serves as the control group to compare against the Pentoxifylline arm in evaluating the potential effect of Pentoxifylline on vascular calcification.
  Interventions: Other: Conventional Medications for Chronic Kidney Disease

INTERVENTIONS:
Drug: Pentoxifylline 400 MG Oral Tablet — Oral tablet, 400 mg, administered twice daily with food for 6 months. To be taken in addition to conventional medications for chronic kidney disease.
  Arms: Pentoxifylline Arm
Other: Conventional Medications for Chronic Kidney Disease — This arm receives conventional medical management for chronic kidney disease (CKD). This includes medications and treatments as deemed necessary and appropriate by the participant's treating physician, according to established clinical guidelines for CKD. These may include, but are not limited to, medications for blood pressure control, management of diabetes, anemia treatment, mineral and bone disorder management, and fluid and electrolyte balance management. The specific medications and treatments are individualized and not dictated by the study protocol, but follow standard clinical practice for CKD.
  Arms: Conventional Medication Group

SUMMARY:
This study is research to find out if the drug pentoxifylline can help prevent or lessen the problem of blood vessel hardening (vascular calcification) in people with chronic kidney disease (CKD). People with CKD are at higher risk for heart problems and blood vessel hardening. Vascular calcification happens when calcium builds up in the blood vessels, making them stiff. Pentoxifylline is a drug that might have helpful effects that could reduce this hardening. In this study, some CKD patients will receive pentoxifylline in addition to their usual medications, while others will only receive their usual medications. The researchers will then compare the amount of vascular calcification in both groups over 6 months to see if pentoxifylline makes a difference. The goal is to learn if pentoxifylline could be a new way to protect the blood vessels of people with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Estimated Glomerular Filtration Rate (eGFR) less than 60 ml/min/1.73 m² and greater than or equal to 15 ml/min/1.73 m².
* Adult patients, age 18 years or older.
* Diagnosis of Chronic Kidney Disease (CKD).
* Willing and able to provide informed consent.

Exclusion Criteria:

* Patients currently undergoing regular hemodialysis.
* History of kidney transplantation or are kidney transplant recipients.
* Pregnant females.
* Patients with a history of coronary artery bypass grafting (CABG).
* Known allergy or contraindication to pentoxifylline.
* Inability to comply with study procedures or attend follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in Agatston Coronary Artery Calcification Score from Baseline to 6 Months | 6 Months
  The primary outcome measure is the change in coronary artery calcification as assessed by the Agatston score, measured from baseline to 6 months after the start of the intervention. Coronary artery calcification will be quantified using computed tomography (CT) scans and analyzed using the Agatston method. A higher Agatston score indicates a greater degree of coronary artery calcification. The change will be calculated as the difference between the Agatston score at 6 months and the Agatston score at baseline.

SECONDARY OUTCOMES:
Change in Estimated Glomerular Filtration Rate (eGFR) from Baseline to 6 Months | 6 Months
  Change in estimated glomerular filtration rate (eGFR) will be assessed from baseline to 6 months. eGFR will be calculated using serum creatinine levels and a standard CKD-EPI equation. eGFR is a measure of kidney function, with lower values indicating poorer kidney function. The change will be calculated as the difference between the eGFR value at 6 months and the eGFR value at baseline.

IPD SHARING:
Plan to Share IPD: Undecided
We are currently undecided about IPD sharing. Factors under consideration include institutional data-sharing policies, ethical considerations related to participant privacy, and the resources required for data anonymization and preparation for sharing. A decision will be made as these factors are further evaluated.

REFERENCES:
- [Background] Leporini C, Pisano A, Russo E, D Arrigo G, de Sarro G, Coppolino G, Bolignano D. Effect of pentoxifylline on renal outcomes in chronic kidney disease patients: A systematic review and meta-analysis. Pharmacol Res. 2016 May;107:315-332. doi: 10.1016/j.phrs.2016.03.001. Epub 2016 Mar 17. PMID 26995301
- [Background] de Morales AM, Goicoechea M, Verde E, Carbayo J, Barbieri D, Delgado A, Verdalles U, de Jose AP, Luno J. Pentoxifylline, progression of chronic kidney disease (CKD) and cardiovascular mortality: long-term follow-up of a randomized clinical trial. J Nephrol. 2019 Aug;32(4):581-587. doi: 10.1007/s40620-019-00607-0. Epub 2019 Apr 4. PMID 30949987
- [Background] Chen J, Budoff MJ, Reilly MP, Yang W, Rosas SE, Rahman M, Zhang X, Roy JA, Lustigova E, Nessel L, Ford V, Raj D, Porter AC, Soliman EZ, Wright JT Jr, Wolf M, He J; CRIC Investigators. Coronary Artery Calcification and Risk of Cardiovascular Disease and Death Among Patients With Chronic Kidney Disease. JAMA Cardiol. 2017 Jun 1;2(6):635-643. doi: 10.1001/jamacardio.2017.0363. PMID 28329057